CLINICAL TRIAL: NCT02109211
Title: Does Altering The Magill Forceps Angle By 45 Degrees Alter Nasal Intubation Time In Pediatric Dental Surgery Patients?
Brief Title: Does Altering Magill Forceps Affect Nasal Intubation Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, William McKay, Faculty, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-250
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Nasal Intubation; Dental Surgery; Pediatrics
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care - Magill forceps (Other): Patients will be intubated, as per standard care, with Magill forceps.
  Interventions: Device: Intubation with Magill forceps
- Altered Magill forceps (Experimental): Patients will be intubated with modified Magill forceps.
  Interventions: Device: Intubation with altered Magill forceps

INTERVENTIONS:
Device: Intubation with Magill forceps
  Arms: Standard care - Magill forceps
Device: Intubation with altered Magill forceps
  Arms: Altered Magill forceps

SUMMARY:
The purpose of this study is to see whether altering the angle of the Magill forceps by 45 degrees will affect nasal intubation time in pediatric dental surgery patients.

The null hypothesis is that their will be no difference between the nasal intubation times of those patients intubated with the conventional Magill forceps and those intubated with the altered Magill forceps.

DETAILED DESCRIPTION:
The Magill forceps (MF) is the instrument of choice for nasal tracheal intubation (NTI). It serves as an aid for inserting the endotracheal tube tip past the vocal cords during NTI. NTI is preferred over oral tracheal intubation (ETT) in certain instances such as pediatric dental surgery. This is because NTI permits excellent access to all intraoral structures while reducing risk of inadvertent displacement of an orotracheal tube. Although there is literature looking at MF design alterations to reduce complications and improve its other uses, there is no literature examining the effect of design alterations on time to successful intubate (TTI). Our study premise is based on the concept that a MF is not ideally structured for the pediatric airway anatomy. Knowing that the larynx is considerably anterior in the pediatric airway, we hypothesized that a + 45° angle change 2cm from the tip of the MF will help align the direction the instrument carrying the endotracheal tube with the anatomic direction of the airway and thus help reduce the TTI.. If a reduction in TTI can be shown it would be of significant benefit and could add another tool for NTI. Even though, the current MF has been satisfactory in its use, this should not deter us from looking for opportunities to improve on the current standard. To test this hypothesis, we will include a hundred participants as part of an open label, controlled, single center, and randomized study in which 50 patients will be intubated with the conventional MF and 50 patients will be intubated with the altered MF. We expect the results to show at least a 5 second reduction in TTI and thus be statistically significant with a p value less than 0.05 for our sample size. Our expected conclusion is that a reduced TTI is clinically beneficially as it will reduce apnea time in the pediatric patients, a population with known physiological limitations in respiratory reserve. This, in turn, could point to a reduction in intra-operative and post-operative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* age 0-15yrs, ASA < or = 2, Mallampati < or = 3, presenting of dental surgery

Exclusion Criteria:

* patients at risk for aspiration, upper airway abnormalities, known difficult airway

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 133 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Time to intubate | Right after measurement
  Having a stopwatch to time how long it takes for the intubator to place initiate direct laryngoscopy until the time of detection of end tidal carbon dioxide on the monitor

SECONDARY OUTCOMES:
Cormack-Lehane glottis view | immediately
  what view is attained through laryngoscopy
Number of attempts to nasal tracheal intubation | once intubation completed
Number of technique failures | once intubation is complete
  To see which other methods of intubation, if any, were needed/used to successfully intubate patient

CONTACTS AND LOCATIONS:
Locations (1):
- Prairieview Surgical Center, Saskatoon, Saskatchewan, Canada